CLINICAL TRIAL: NCT04460612
Title: A Pilot Study of the Impact of Passive, Garment-based Infrared Therapy on Oxygenation in the Feet and Lower Legs of Patients With Diabetes
Brief Title: Infrared Wraps Effect on Oxygenation of Diabetics Arm, Feet and Lower Leg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: CIRCUFIBER, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000027079
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Double Blind Randomized Placebo Controlled using the patients as their own controls. Patients will be randomized to receive either placebo wraps or the infrared wraps and then crossover to the alternative wrap.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Infrared wraps will be compared to non-infrared placebo wraps which are identical in appearance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Sock (Placebo Comparator): Placebo Socks will be placed on participants feet either first or second for 60 minutes
  Interventions: Device: Active IR sock; Other: Placebo socks
- Active IR Sock (Active Comparator): Active IR socks will be placed on participants feet either first or second
  Interventions: Device: Active IR sock; Other: Placebo socks

INTERVENTIONS:
Device: Active IR sock — Subjects will be wearing the infrared socks for 60 minutes
  Other Names: Infrared sock
Other: Placebo socks — Placebo Socks will be placed on participants feet first for 60 minute

SUMMARY:
This study seeks to prove that wraps manufactured with infrared textile are capable of augmenting peripheral circulation in the lower legs, arm and feet of participants with Diabetes Mellitus. Infrared is currently used in saunas and various textiles as general wellness products that purport to improve various health conditions and augment microcirculation. This study is intended to investigate specifically whether wraps capable of harnessing infrared energy can improve oxygenation in the feet, arms and lower legs of diabetics using noninvasive transcutaneous oximetry to do so.

DETAILED DESCRIPTION:
Infrared energy is a type of electromagnetic energy that is invisible, and is further subdivided into three subsets based on wavelength. Far infrared (FIR or IR-C) is a subset of energy in the infrared spectrum that is thought to transfer energy in the form of heat, perceived by thermoreceptors in the skin as radiant heat. FIR is thought to be both absorbed by the human body but is also emitted in the 3-50 micron range, with a peak output at 9.4 micron. The range of far infrared varies depending on which source is referenced but is generally felt to start at 3 to 5 microns. The use of FIR has been studied in various circumstances and thought to improve various biological functions via FIR heat lamps, saunas, ray devices and FIR emitting ceramics and fabrics. There are no short-term or long-term safety issues that have arisen in any studies thus far. As noted in the 2006 statement of the ICNIRP (International Commission on Non-Ionizing Radiation Protection), "…the contribution made by the IR-C spectral region (3-1,000 micron) is normally of no practical concern from a health hazard standpoint." FIR has been shown to increase blood flow in forearms, and access flow and survival of arteriovenous fistula in hemodialysis patients. An unpublished study, by McClue, reported an apparent increase in pedal circulation of approximately 10% using transcutaneous oxygen monitoring in healthy subjects wearing socks infiltrated with FIR emitting textiles. The mechanism of improving circulation is not entirely elucidated, however recent work suggests a role of increasing endothelial nitric oxide synthase, nitric oxide production and modulating profiles of circulating miRNAs (mircoRNA, small noncoding RNAs of ∼22nt in length which are involved in the regulation of gene expression at the posttranscriptional level).

Type 2 Diabetes prevalence has increased significantly over the past decade, with estimates from 2015 of 26 million Americans diagnosed and predicted to increase to 32 million by 2020. Both Type 1 and Type 2 Diabetes is well known to increase the risk of nontraumatic lower extremity amputation by, amongst other factors, impairing circulation to the feet through both peripheral arterial disease and microvascular dysfunction.

Noninvasive transcutaneous oximetry measurements of the leg have been validated as a valuable tool in assessing lower extremity circulation in both normal subjects and diabetic individuals.

This trial seeks to prove that exposure to IR, through the use of newly developed socks (wraps here with same material) that contain thermoreactive particles woven into textile, which both emit IR and reflect the IR back from the body, can augment circulation in the feet, arms and lower legs of diabetic subjects. Noninvasive transcutaneous oximetry will be used as the assessment modality. If this study confirms this hypothesis, future studies may be planned to determine if the use of a IR-containing textile can prevent new ulcers from forming in high risk patients and perhaps even speed the healing of prevalent foot ulcers.

Subjects will be recruited from both primary care and specialty medical offices who carry a diagnosis of Diabetes Mellitus, will be between the ages of 18 to 80 and will act as their own controls. The goal will be to enroll a minimum of one hundred (100) patients who will be evaluated noninvasively with transcutaneous oxygen measurements using Radiometer TCM (PeriFlux 5000) supplied by Radiometer America, Inc. Upon screening and after signing informed consent, patients will have ankle brachial index (ABI) measurements performed on both legs to exclude those who have severe peripheral arterial disease (ABI index or 0.4 or lower). Upon arrival on study day, subjects will have both feet evaluated by a registered nurse (RN), to ensure there are no signs of infection, active foot ulcers, or other open wounds. If there is any such evidence, the patients will be excluded from the trial and sent for further evaluation and treatment according to standard of care by their primary care clinicians or podiatrists.

Subjects will be placed on an exam table reclined at a 120-degree angle with legs extended and supported by leg rest. The TCPO2 machine will have been turned on prior to patient arrival for calibration. If necessary, any hair on the subject's foot or leg will be removed in the area of fixation ring application by a disposable razor. The subject will then have up to 3 fixation rings attached, used for measuring TCPO2, placed on the lower leg and foot. The fixation rings will be further secured around the circumference with medical tape, approximately 1 inch by 0.5 inch per piece to further enhance the seal. In a double blind fashion, subjects will be randomized to have either placebo or IR wraps placed in a sequential way. The wrap will be placed over the foot, arm and lower leg covering the fixation rings. Three drops of contact solution will be placed inside each fixation ring, followed by attachment of the electrodes. There will then be a 30 minute rest/stabilization period allowing for the TCPO2 to stabilize (stabilization phase).

The wraps will then be gently applied to the arm, feet and leg, while being careful not to disturb the fixation rings. The placebo wraps are identical in all ways to the study wrap, with the exception that the placebo wraps do not contain the proprietary thermoreactive minerals woven into the fabric. The active phase will then commence and continue for 60 minutes, with TCPO2 measurements taking place continuously and recorded at least every 10 minutes. At the end of the 60-minute study period, the leads will be removed, followed by the wraps. The fixation rings are not removed, however. The TCPO2 machine should be recalibrated after the leads are returned to the holding chamber, prior to the second half of the trial using the other wraps (either IR or placebo, whichever was not used in first session). There will then be a 10-minute break period, subjects will be allowed to use the restroom and may place loose foot coverings over their feet for ambulation. Following the subjects return to the exam table, the same above protocol will be followed, with 30 minutes of rest/stabilization after the leads are placed back on for the baseline readings prior to wrap placement. Repeat TCPO2 measurements will be obtained according to the same schedule as indicated above. Activity will be restricted during the active and stabilization phase of the protocol. Patients will be encouraged to void prior to initiation of each half of the protocol. However, should subjects have to use the bathroom during one of the active phases, the rest and stabilization phase will restart at time zero following the bathroom break and reattachment of the TCPO2 sensors. At the completion of the study, the leads and fixation rings will be removed and subjects will return placebo and study socks to the appropriate personnel.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Type 1 or Type 2 Diabetes Mellitus between the ages of 18 and 80 years old.

Exclusion Criteria:

* Chronic kidney disease treated by dialysis or those with a eGFR<30 mL/min/1.73m2
* Alcohol or any illicit substance abuse
* Use of systemic corticosteroids within previous 3 months
* Has ever received immunosuppressive agents
* Has ever undergone radiation therapy
* Has ever used cytotoxic agents
* Pregnant, breast-feeding or attempting to become pregnant
* History of known peripheral arterial disease or lower extremity amputation
* Any neurologic disease or other condition preventing normal ambulation
* History of significant trauma to the lower extremities, major orthopedic or neurological damage to the lower extremities
* History of saphenous venous graft harvesting
* Ankle-Brachial Index of 0.40 or lower
* Any ulcer or open wound on the lower extremities
* Inability to lie flat for up to 90 minutes at a time
* Any symptoms within past 21 days of cough, fever, sore throat, chills, body aches, shortness of breath, loss of smell, loss of taste, fever at or greater than 100 degrees Fahrenheit
* COVID positive nasal swab within past 21 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Change in oxygenation of feet and lower legs | 60 minutes
  Transcutaneous oxygen measurements will be compared between placebo and active IR sock

CONTACTS AND LOCATIONS:
Overall Officials: Adam B Mayerson, M.D., Principal Investigator — Yale University
Locations (1):
- Endocrine Associates Of Connecticut, Hamden, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share IPD.

REFERENCES:
- [Background] Shui S, Wang X, Chiang JY, Zheng L. Far-infrared therapy for cardiovascular, autoimmune, and other chronic health problems: A systematic review. Exp Biol Med (Maywood). 2015 Oct;240(10):1257-65. doi: 10.1177/1535370215573391. Epub 2015 Feb 25. PMID 25716016 (Retraction: PMID 32686476 Exp Biol Med (Maywood). 2020 Aug;245(14):NP1)
- [Background] Vatansever F, Hamblin MR. Far infrared radiation (FIR): its biological effects and medical applications. Photonics Lasers Med. 2012 Nov 1;4:255-266. doi: 10.1515/plm-2012-0034. PMID 23833705
- [Background] Lin CC, Chang CF, Lai MY, Chen TW, Lee PC, Yang WC. Far-infrared therapy: a novel treatment to improve access blood flow and unassisted patency of arteriovenous fistula in hemodialysis patients. J Am Soc Nephrol. 2007 Mar;18(3):985-92. doi: 10.1681/ASN.2006050534. Epub 2007 Jan 31. PMID 17267744
- [Background] Ise N, Katsuura T, Kikuchi Y, Miwa E. Effect of far-infrared radiation on forearm skin blood flow. Ann Physiol Anthropol. 1987 Jan;6(1):31-2. doi: 10.2114/ahs1983.6.31. No abstract available. PMID 3675759
- [Background] Rowley WR, Bezold C, Arikan Y, Byrne E, Krohe S. Diabetes 2030: Insights from Yesterday, Today, and Future Trends. Popul Health Manag. 2017 Feb;20(1):6-12. doi: 10.1089/pop.2015.0181. Epub 2016 Apr 28. PMID 27124621
- [Background] Geiss LS, Li Y, Hora I, Albright A, Rolka D, Gregg EW. Resurgence of Diabetes-Related Nontraumatic Lower-Extremity Amputation in the Young and Middle-Aged Adult U.S. Population. Diabetes Care. 2019 Jan;42(1):50-54. doi: 10.2337/dc18-1380. Epub 2018 Nov 8. PMID 30409811
- [Background] Trinks TP, Blake DF, Young DA, Thistlethwaite K, Vangaveti VN. Transcutaneous oximetry measurements of the leg: comparing different measuring equipment and establishing values in healthy young adults. Diving Hyperb Med. 2017 Jun;47(2):82-87. doi: 10.28920/dhm47.2.82-87. PMID 28641320
- [Background] Zimny S, Dessel F, Ehren M, Pfohl M, Schatz H. Early detection of microcirculatory impairment in diabetic patients with foot at risk. Diabetes Care. 2001 Oct;24(10):1810-4. doi: 10.2337/diacare.24.10.1810. PMID 11574447
- [Background] International Commission on Non-Ionizing Radiation Protection (ICNIRP). ICNIRP statement on far infrared radiation exposure. Health Phys. 2006 Dec;91(6):630-45. doi: 10.1097/01.HP.0000240533.50224.65. No abstract available. PMID 17099407
- [Background] McClue G, Celliant Study of Thirteen (13) Healthy Subjects. 2005 (unpublished) https://celliant.com/wp-content/uploads/2020/04/Celliant-Published-Studies-Compilation-of-Clinical-Technical-and-Physical-Trials-April-2020-min.pdf